CLINICAL TRIAL: NCT02829879
Title: Comparison of the Clinical Effectiveness of 8% Arginine/1450 Ppm Sodium Monofluorophosphate Versus 5% Potassium Nitrate/2500 Ppm Sodium Fluoride in Dentin Hypersensitivity Therapy: A Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Arginin and Potassium Nitrate Dentifrices in Dentin Hypersensitivity Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Patricia Hernández-Ríos, Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIOUCh 13-103
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Dentin Sensitivity
Keywords: Dentin Sensitivity; Arginin; Potassium Nitrate; Dentifrice; RCT
MeSH Terms: conditions — Dentin Sensitivity | interventions — Arginine; potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- arginine (Experimental): 25 volunteers with dentin sensitivity
  Interventions: Drug: 8% arginine/1450ppm sodium monofluorophosphate dentifrice
- potassium nitrate (Active Comparator): 25 volunteers with dentin sensitivity
  Interventions: Drug: 5% potassium nitrate/2500ppm sodium fluoride dentifrice

INTERVENTIONS:
Drug: 8% arginine/1450ppm sodium monofluorophosphate dentifrice
  Arms: arginine
Drug: 5% potassium nitrate/2500ppm sodium fluoride dentifrice
  Arms: potassium nitrate

SUMMARY:
Introduction: Dentin hypersensitivity (DH) could be defined as a brief and sharp pain in response to thermical, chemical, tactile and osmotic stimuli, which cannot be attributed to any dental condition or pathology. Multiple therapies for the treatment of DH have been studied, including equivocal evidence about the efficacy of potassium nitrate salts and recent investigations a promising new 8% Arginin dentifrice.

Aim: The aim of this study is to compare the clinical effectiveness of 8% arginine/1450ppm sodium monofluorophosphate (D1) and 5% potassium nitrate/2500ppm sodium fluoride (D2) dentifrices in the treatment of dentin hypersensitivity.

Methods: Parallel-design, double-masked, randomized controlled clinical trial. Fifty healthy volunteers aged 18 to 70 years who attend at the Faculty of Dentistry , University of Chile, with DH and a visual analog scale (VAS) score ≥4 at least in two anterior and/or premolar teeth, will be selected and randomized into two treatment groups: T1 (n=25): 8% arginine/1450 ppm sodium monofluorophosphate dentifrice (D1); and T2 (n=25): 5% potassium nitrate/2500 ppm sodium fluoride dentifrice (D2). Environmental, dietary and oral hygiene habits will be recorded in a clinical chart, while O´Leary plaque index and dentin hypersensitivity (DH) measurements will be clinically assessed, at baseline, 4 and 8 weeks. DH will be evaluated through the mean VAS value in response to evaporative and thermal stimuli at baseline, 4 and 8 week follow-up. The data will be analysed through Stata® V11 program.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Dentin sensitivity in at least 2 teeth (incisors, cuspids and/or bicuspids) with a VAS score ≥4
* Good general health

Exclusion Criteria:

* Defective or extensive restorations, deep dental caries, pulpitis, chipped teeth,
* Bridgework, dentures or crowned teeth that could interfere with the evaluation of hypersensitivity
* Pregnancy or lactation
* Ongoing treatment with anti-inflammatory or sedative drugs
* Systemic conditions that are etiologic or predisposing to dentine hypersensitivity, like chronic acid regurgitation
* Ongoing periodontal therapy or periodontal surgery in the preceding 3 months
* Allergic responses to the dentifrices
* Hypersensitivity treatment in the preceding 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Differences in mean VAS score per subject | Baseline, 4 and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University of Chile, Santiago, Santiago Metropolitan, Chile